CLINICAL TRIAL: NCT03500497
Title: The Change in RetHe - Levels Perioperatively in a Cohort of Colorectal Surgery Patient: it's Role in Perioperative Hemoglobin Optimization
Brief Title: The Change in RetHe - Levels Perioperatively in a Cohort of Colorectal Surgery Patient
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RACEmumc
Record Dates: First submitted 2018-02-14; First posted 2018-04-18 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Anemia; Colorectal Surgery; Perioperative
Keywords: reticulocyte hemoglobin content (RetHe); perioperative; colorectal surgery; anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Diagnostic Test: RetHe measurement (Sysmex) — RetHe measurement is done from blood samples gained during standard patient care perioperatively

SUMMARY:
During a period of a year, reticulocyte hemoglobin content (RetHe) measurements (Sysmex) are done out of blood samples taken on several occasions during normal patient care:

1. preoperatively at the surgical or anesthetic outpatient visit
2. on admission or pre- induction of anesthesia
3. postoperatively at the postanesthetic care unit
4. on day 3 postoperatively
5. on day 5 postoperatively

Additionally a Quality of Life (QoL) questionnaire will be taken from the participants before surgery and 30 days after surgery to evaluate the course of QoL perioperatively.

DETAILED DESCRIPTION:
Study design An explorative, prospective cohort study of patients undergoing colorectal surgery in the Maastricht University Medical Center (MUMC) with a follow-up time of 30 days postoperatively.

A quality of life questionnaire (EQ-5D) will be administered on admission and 30 days postoperatively.

Origin of data Medical file of patients (SAP, PDMS) Database Study data are anonymous information, which cannot be tracked to the patient according to wet bescherming persoonsgegevens (WBP) and wet op geneeskundige behandelingsovereenkomst (WGBO). These will be stored at Castor Electronic Data Capture (EDC), secure online data collection for medical research), that embraces Good Clinical Practice (GPC) guidelines. For the analysis, anonymized data will be exported to Statistical Package for the Social Sciences (SPSS).

Preoperative anemia in the colorectal surgical population is a common and independent risk factor of perioperative morbidity and mortality. The detection, diagnostic and treatment of anemia are therefore a multidisciplinary obligation in the optimization of patient care.

In the perioperative setting anemia can be divided into three categories:

* Pre-existing anemia prior to surgery (blood loss, chronic and acute inflammatory response, increased destruction (haemolysis), chemotherapy)
* Anemia caused by the surgical intervention (blood loss, acute inflammatory response, increased destruction)
* Anemia due to iatrogenic causes (blood sampling, haemodilution)

Adequate diagnostic is needed to determine anemia in the perioperative setting in order to guide appropriate further therapy.

Preoperative diagnostic approaches have recently been implemented to direct the treatment of pre-existing anemia with the intention to optimize preoperative hemoglobin levels. Laboratory evaluation is based on measurements of ferritin, transferrin saturation (TfS), C-reactive protein (CRP) and renal function to screen for the underlying cause of anemia. One compelling component of the preoperative augmentation of haemoglobin level is intravenous iron administration in case of absolute or functional iron deficiency.

Unfortunately, the laboratory diagnostic of iron status is limited due to the interaction of inflammatory response with the markers (ferritin, TfS). As the main goal of therapy is haemoglobin optimization it seems appropriate to use erythropoietic parameters to assess the adequacy of iron therapy. The hemoglobin content of the reticulocyte (RetHe), which describes the erythropoietic responsiveness to iron therapy at the level of erythrocytes precursors, has been shown to be a sensitive and rapid marker. Since reticulocytes have a more rapid turnover in circulation than mature red cells (1-2 vs 120 days), it is hypothesized that the assessment of RetHe can mirror responsiveness to therapy within the perioperative setting in a more timely manner. Moreover the course of perioperative RetHe has not been examined and the aim of this study is to assess the differences in RetHe between the participants and during their time of admission.

Therefore this parameter could be useful in the perioperative period to further guide adequate management.

Another aspect that we would like to track is the influence of iron deficiency +/- anemia on quality of life (QoL) in this patient group. While some studies show a strong relationship between iron deficiency anemia on QoL in patients with cancer or ischemic bowel disease, the overall effect in the perioperative setting remains unproven.

In our setting we experience a very variable time frame for preoperative patient optimization in relation with organizational issues and urgency of surgery. The required time period from diagnosis to actual operation for elective procedures is nominated to be maximal 3 weeks.

To give all patients the chance to optimize anemia preoperatively or support postoperative erythropoetic activity, we have determined in a multidisciplinary advisory to use intravenous iron as soon as possible after diagnosis, including the day of operation.

To our knowledge, RetHe has not been assessed as a progression parameter for iron therapy in clinical setting within that patient group. Cut off values are validated. Because reticulocyte parameters change within 24 -48 hours, we chose RetHe rather than hemoglobin (Hb) as biochemical marker of bone marrow activity.

Clinical practice During a period of a year all participants scheduled for colorectal surgery will be included. Registration of hematological parameters includes the hemoglobin concentration, mean cell volume (MCV), mean corpuscular hemoglobin concentration (MCHC) and RetHe. The iron status is recorded by ferritin and transferrin saturation preoperatively. CRP and renal function tests are followed to differentiate the cause of anemia and to guide perioperative management. Interventions, which interact with the hemoglobin level will be registered. All laboratory investigations are standardized care in our institution. The RetHe measurement can be retrieved out of the same blood sample used in standard care. Beyond that also kind and length of operation and postoperative morbidity and mortality are of interest.

Data collection:

A study-specific internet-based case record form will be used to register specific study data and complications (Castor EDC). Assessment of postoperative complications are scored according to the Calvien-Dindo classification. All of the study parameters are part of the routine medical record of surgical patients and can be derived from electronic patient files.

The only hematological diagnostic which are beyond our current standardized care is RetHe, which can be measured in the same blood sample as taken for Hb measurement. No additional blood sampling is needed.

The Functional Assessment of Cancer Therapy - Anemia (FACT-An) questionnaire will be administered preoperatively and 30 days postoperatively on paper or digital based on participant preference. Completed questionnaires on paper will be entered in Castor EDC manually.

Statistical analysis The prevalence of preoperative anemia and perioperative complications will be reported as frequencies and percentages, accompanied by a measure of precision.The variance of RetHe values between participants will be computed. We will plot figures to explore the average RetHe and Hb values from baseline to postoperatively. Using an independent t-test, we will test the difference in preoperative RetHe values between anemic patients and those who are not anemic. Hematological parameters as well as inflammatory marker and organ function tests will be analyzed in view of iron supplementation.

A cost assessment for the use of intravenous iron, postoperative complications and hospital stay will be included in the final study analysis.

Patient benefit For the patients who will participate in this current study there are no direct benefits. Nor is there any harm or even increased burden for them. However, for future patients results form this study could prove very beneficial in terms of individualized anemia optimization perioperatively. This has the potential to improve postoperative outcome and the QoL of the patients.

Data management Data will be handled confidentially. Participants will be given a random study identification code that is not based on the participants' birth date or initials. One way coding using ascending numbers will be used. Access to the coding system is only granted to the investigators. Additionally we will record anonymous participant data, which are registered routinely throughout hospital admission, for audit purposes to complete our data.

The blood samples of the participants will be managed as it is required for standard patient care, but in agreement with the participant, they will be stored until the study is completed, so that additional measurements can be done. As RetHe is not a standardized parameter in clinical care, its comparison with the current standard assay (ferritin and TfS) may be warranted as part of this investigation to amplify findings.

The data management system Castor EDC will be used for electronic Case Report Forms (eCRFs) and storage of the study data. Castor EDC is fully compliant with GPC guidelines on data safety. After the study, all data will be kept for 15 years for verification purposes.

Publication policy Both positive and negative results of this study will be disclosed unreservedly through publication in peer-reviewed scientific journals.

Informed consent As the Human Subjects study protocol may be assessed as non-WMO (wet medish wetenschappelijk onderzoek) research, written informed consent will be gained from the prospective cohort (see appendix). No historic cohort needs to be analyzed as the study is merely prospective.

The participants will be first informed about the study when referred for surgery by the treating doctor. They will receive the patient information sheet and will be given time to consider their participation. Usually more than a week, but minimally one day for elective procedures. In case of emergency procedures, informed consent will be asked at the same time as anesthetic consent. The investigator is responsible for timely information about the study and the obtainment of consent.

Data, which will be collected, are strictly not identifiable personal information and collection, storage and analysis will be according to the Code of Conduct (Gedragscode Gezondheidsonderzoek, article 3).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥ 18 years) scheduled for colorectal surgical operations (laparoscopic and open procedures)

Exclusion Criteria:

* emergency surgery
* minors and incapacitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elective colorectal surgery patients (cancer surgery, inflammatory disease, other pathologies needing elective intestinal surgery)
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Change of RetHe measurement | From baseline to 60 days postoperatively
  To assess the change of RetHe measurement from baseline (preoperative assessment) to different points in time in standard care (i.e. RetHe measurement at day of admission, direct postoperatively and day 3 and 5 postoperatively)

SECONDARY OUTCOMES:
Relation of RetHe to standard iron status measurements | 1 year
  In case of relevant RetHe aberrations those will be compared to the standard iron status measurements (i.e. transferrin saturation and ferritin)
Perioperative complications | Days of admission
  The complications will be scaled according to the Calvien-Dindo classification
Quality of life measurement preoperatively and 30-days postoperatively | From baseline to 30-days postoperatively
  Validated quality of life patient questionnaire (i.e. FACT-An) is asked from the preoperatively and 30-days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia S Mueller, Dr, Principal Investigator — MUMC Maastricht
Locations (1):
- MUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be handled confidentially. Patients included in the study will be given a random study identification code that is not based on the patients' birth date or initials. One way coding using ascending numbers will be used. Access to the coding system is only granted to the investigators.

REFERENCES:
- [Background] Aapro M, Osterborg A, Gascon P, Ludwig H, Beguin Y. Prevalence and management of cancer-related anaemia, iron deficiency and the specific role of i.v. iron. Ann Oncol. 2012 Aug;23(8):1954-1962. doi: 10.1093/annonc/mds112. Epub 2012 May 9. PMID 22575608
- [Background] Archer NM, Brugnara C. Diagnosis of iron-deficient states. Crit Rev Clin Lab Sci. 2015;52(5):256-72. doi: 10.3109/10408363.2015.1038744. Epub 2015 Aug 14. PMID 26292073
- [Background] Clevenger B, Richards T. Pre-operative anaemia. Anaesthesia. 2015 Jan;70 Suppl 1:20-8, e6-8. doi: 10.1111/anae.12918. PMID 25440391
- [Background] Froessler B, Palm P, Weber I, Hodyl NA, Singh R, Murphy EM. The Important Role for Intravenous Iron in Perioperative Patient Blood Management in Major Abdominal Surgery: A Randomized Controlled Trial. Ann Surg. 2016 Jul;264(1):41-6. doi: 10.1097/SLA.0000000000001646. PMID 26817624
- [Background] Gozzard D. When is high-dose intravenous iron repletion needed? Assessing new treatment options. Drug Des Devel Ther. 2011 Jan 20;5:51-60. doi: 10.2147/DDDT.S15817. PMID 21340038
- [Background] Herrera-deGuise C, Casellas F, Robles V, Navarro E, Borruel N. Iron Deficiency in the Absence of Anemia Impairs the Perception of Health-Related Quality of Life of Patients with Inflammatory Bowel Disease. Inflamm Bowel Dis. 2016 Jun;22(6):1450-5. doi: 10.1097/MIB.0000000000000768. PMID 27057682
- [Background] Jans O, Bandholm T, Kurbegovic S, Solgaard S, Kjaersgaard-Andersen P, Johansson PI, Kehlet H; Lundbeck Foundation Centre for Fast-Track Hip and Knee Replacement Collaborative Group. Postoperative anemia and early functional outcomes after fast-track hip arthroplasty: a prospective cohort study. Transfusion. 2016 Apr;56(4):917-25. doi: 10.1111/trf.13508. Epub 2016 Mar 4. PMID 26945552
- [Background] Kanuri G, Sawhney R, Varghese J, Britto M, Shet A. Iron Deficiency Anemia Coexists with Cancer Related Anemia and Adversely Impacts Quality of Life. PLoS One. 2016 Sep 28;11(9):e0163817. doi: 10.1371/journal.pone.0163817. eCollection 2016. PMID 27682226
- [Background] Keeler BD, Mishra A, Stavrou CL, Beeby S, Simpson JA, Acheson AG. A cohort investigation of anaemia, treatment and the use of allogeneic blood transfusion in colorectal cancer surgery. Ann Med Surg (Lond). 2015 Dec 22;6:6-11. doi: 10.1016/j.amsu.2015.12.052. eCollection 2016 Mar. PMID 26909150
- [Background] Beale AL, Penney MD, Allison MC. The prevalence of iron deficiency among patients presenting with colorectal cancer. Colorectal Dis. 2005 Jul;7(4):398-402. doi: 10.1111/j.1463-1318.2005.00789.x. PMID 15932566
- [Background] Mast AE, Blinder MA, Dietzen DJ. Reticulocyte hemoglobin content. Am J Hematol. 2008 Apr;83(4):307-10. doi: 10.1002/ajh.21090. PMID 18027835
- [Background] Mouysset JL, Freier B, van den Bosch J, Levache CB, Bols A, Tessen HW, Belton L, Bohac GC, Terwey JH, Tonini G. Hemoglobin levels and quality of life in patients with symptomatic chemotherapy-induced anemia: the eAQUA study. Cancer Manag Res. 2016 Jan 21;8:1-10. doi: 10.2147/CMAR.S88110. eCollection 2016. PMID 26855598
- [Background] Musallam KM, Tamim HM, Richards T, Spahn DR, Rosendaal FR, Habbal A, Khreiss M, Dahdaleh FS, Khavandi K, Sfeir PM, Soweid A, Hoballah JJ, Taher AT, Jamali FR. Preoperative anaemia and postoperative outcomes in non-cardiac surgery: a retrospective cohort study. Lancet. 2011 Oct 15;378(9800):1396-407. doi: 10.1016/S0140-6736(11)61381-0. Epub 2011 Oct 5. PMID 21982521
- [Background] So-Osman C, Nelissen R, Brand R, Brand A, Stiggelbout AM. Postoperative anemia after joint replacement surgery is not related to quality of life during the first two weeks postoperatively. Transfusion. 2011 Jan;51(1):71-81. doi: 10.1111/j.1537-2995.2010.02784.x. PMID 20663113
- [Background] Thomas DW, Hinchliffe RF, Briggs C, Macdougall IC, Littlewood T, Cavill I; British Committee for Standards in Haematology. Guideline for the laboratory diagnosis of functional iron deficiency. Br J Haematol. 2013 Jun;161(5):639-648. doi: 10.1111/bjh.12311. Epub 2013 Apr 10. No abstract available. PMID 23573815
- [Background] Urrechaga E, Borque L, Escanero JF. Biomarkers of hypochromia: the contemporary assessment of iron status and erythropoiesis. Biomed Res Int. 2013;2013:603786. doi: 10.1155/2013/603786. Epub 2013 Feb 28. PMID 23555091